CLINICAL TRIAL: NCT03260777
Title: Relevance of Trichoscopy in Differential Diagnosis of Focal Non-cicatricial Alopecia in Children
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohamed, Principle Investigator, Assiut University
Other Study IDs: ROTIDDOFNCAIC
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Focal Non-cicatricial Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- children with Alopecia Areata
  Interventions: Device: Trichoscopy
- children with tinea capitis
  Interventions: Device: Trichoscopy
- children with trichotillomania
  Interventions: Device: Trichoscopy
- children with tractional alopecia
  Interventions: Device: Trichoscopy

INTERVENTIONS:
Device: Trichoscopy — Trichoscopy (hair and scalp dermoscopy) is a noninvasive diagnostic tool that allows the recognition of morphologic structures not visible by the naked eye Structures which may be visualized by trichoscopy include hair shafts of different types, the number of hairs in one pilosebaceous unit, hair follicle openings (dots), the peri and interfollicular areas and the vasculature.

SUMMARY:
Alopecia is a common, distressing condition that is sometimes difficult to diagnose and treat.

Losing hair is not usually health threatening; it can scar a young child's vulnerable self-esteem by causing immense psychological and emotional stress, not only to the patient, but also to the concerned parents and siblings; so the cause of hair loss should be diagnosed and treated early to overcome the resulting problems.

DETAILED DESCRIPTION:
The majority of alopecia in children is presented as patchy alopecia, which is most commonly diagnosed as alopecia areata. However, other causes of patchy alopecia such as tinea capitis, trichotillomania, temporal triangular alopecia (TTA), nevus sebaceous and aplasia cutis congenita (ACC) can be easily missed.

Trichoscopy (hair and scalp dermoscopy) is a non-invasive diagnostic tool that allows the recognition of morphologic structures not visible by the naked eye.

Trichoscopy allows visualization of hair shafts at high magnification and performing measurements, such as hair shaft thickness, without the need of removing hair for diagnostic purposes. It also allows in vivo visualization of the epidermal portion of hair follicles and perifollicular epidermis.

The advantages of trichoscopy in evaluating hair loss in children are numerous, as it is a fast in-office technique , non-invasive, inexpensive, and painless , and therefore it will be accepted by children and their parents.

Tinea capitis and alopecia areata are considered to be the most common causes of hairless patches of the scalp in pediatrics. Tinea capitis especially non-scaly type may have the same clinical appearance of alopecia areata, so trichoscopy has recently become a useful diagnostic tool for alopecia areata and tinea capitis, especially in doubtful cases as lab investigations like fungal culture or biopsy may take several weeks.

ELIGIBILITY:
Inclusion Criteria:

-age from 3-18 years of both sexes with focal non-cicatricial alopecia.(1-5 patches of alopecia)

Exclusion Criteria:

1. Patients who will not consent.
2. uncooperative children.
3. patients with active secondary bacterial infection in the alopecic patch.
4. patients with any concomitant dermatological diseases.
5. history of using any topical(1 month) or systemic treatment (3 month) for tinea capitis or alopecia areata prior to the study,
6. cicatricial alopecia.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 Patients with focal non-cicatricial alopecia will be recruited from the outpatient clinic of Dermatology , Venereology and Andrology department at Assiut University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the common trichoscopic findings in diagnosis of clinically difficult cases of focal non-cicatricial alopecia in children. | 2017-2018
  Characteristic trichoscopic findings will be searched for in each case such as (exclamation mark hairs, yellow and black dots) for alopecia areata. Flame hairs, tulip hairs, coiled hairs, hook hairs, v-sign and irregularly broken hairs for trichotillomania.Findings for tinea capitis (comma hairs, zigzag hairs, corkscrew hairs and block hairs).Coiled irregularly broken hairs and hair casts for tractional alopecia.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Universuty, Asyut, Egypt

REFERENCES:
- [Background] Lencastre A, Tosti A. Role of trichoscopy in children's scalp and hair disorders. Pediatr Dermatol. 2013 Nov-Dec;30(6):674-82. doi: 10.1111/pde.12173. Epub 2013 Aug 13. PMID 23937326
- [Background] Miteva M, Tosti A. Hair and scalp dermatoscopy. J Am Acad Dermatol. 2012 Nov;67(5):1040-8. doi: 10.1016/j.jaad.2012.02.013. Epub 2012 Mar 8. PMID 22405573
- [Background] Sarifakioglu E, Yilmaz AE, Gorpelioglu C, Orun E. Prevalence of scalp disorders and hair loss in children. Cutis. 2012 Nov;90(5):225-9. PMID 23270190
- [Background] Rakowska A. Trichoscopy (hair and scalp videodermoscopy) in the healthy female. Method standardization and norms for measurable parameters. J Dermatol Case Rep. 2009 Apr 5;3(1):14-9. doi: 10.3315/jdcr.2008.1021. PMID 21886722
- [Background] Hillmann K, Blume-Peytavi U. Diagnosis of hair disorders. Semin Cutan Med Surg. 2009 Mar;28(1):33-8. doi: 10.1016/j.sder.2008.12.005. PMID 19341940